CLINICAL TRIAL: NCT02207764
Title: Reiki as a Complementary Therapy: A Pilot Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: competing priorities at the organization
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: J1358; IRB00026755 (Other: JHMIRB)
Record Dates: First submitted 2014-07-29; First posted 2014-08-04 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-07

CONDITIONS: Hematologic Malignancy
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Therapeutic Touch

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Reiki Intervention (Experimental): Each study participant in the intervention group will receive one Reiki intervention by a registered nurse trained in Advanced Level Reiki through the Usui Shiki Ryoho method.
  Interventions: Behavioral: Reiki
- nursing presence control (No Intervention): Each patient in the control group will receive usual care including the study nurse presence for the 15-minute period.

INTERVENTIONS:
Behavioral: Reiki — Each study participant in the intervention group will receive one Reiki intervention by a registered nurse trained in Advanced Level Reiki through the Usui Shiki Ryoho method.
  Arms: Reiki Intervention

SUMMARY:
This research is being done to test whether a complementary intervention, Reiki therapy, can provide added benefits to the standard patient care. Reiki is method for stress reduction that uses hand positions over and/or on the body to help people relax.

We are studying the effect of a 15-minute Reiki application compared to an intervention of nursing presence without Reiki. We hope to find if Reiki can assist in relieving stress, and improving patient outcomes. In the future we would like to offer complementary interventions as an adjunct to our standard care for patients.

DETAILED DESCRIPTION:
This pilot study is designed to test if a complementary therapy, Reiki, has an effect on physiological and subjective measures of stress. This is a 2-arm randomized pilot study of the use of Reiki therapy prior to a stressful event with a convenience sample of 40 participants who are newly diagnosed hematologic malignancy patients on the inpatient service who will experience bone marrow aspirate post induction chemotherapy. Reiki therapy is a non-invasive complementary therapy that can be used in addition to the standard of care. The intervention group will receive a 15-minute Reiki session and the control group will receive 15 minutes of nursing presence. Each study arm includes a brief item questionnaire to rank subjective measures of pain, anxiety, and energy; saliva biological markers related to stress-reduction; and measures of blood pressure, heart rate, and respirations. The intervention group will receive a 15-minute intervention performed on the inpatient unit prior to the bone marrow aspirate procedure. Data will be collected from patients both before and after the intervention and before and after the bone marrow aspirate. We will collect saliva samples from the control group and baseline data including subjective measures of pain, anxiety and energy and measures of blood pressure, heart rate, and respirations. The study nurse will maintain presence in the control participant's room for 15-minutes after the initial measures.

Our research hypothesis is that there will be a change in the response to one or more parameters of physiological or subjective measures for those patients receiving a Reiki intervention when compared to those receiving standard of care plus the nurse presence in room.

The null hypothesis is there will be no difference in response between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 and older admitted to hospital
* Speak English
* Able to give consent will be included.

Exclusion Criteria:

* Patients who are under 18
* Non-English speaking
* Unable to consent
* Pregnant women
* Unwilling to join the study will be excluded
* Intensive Care Unit (ICU) patients and those patients scheduled to receive conscious sedation will be excluded.
* Each patient may join the pilot study only once

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
stress level: patient report | baseline: prior to Reiki intervention
  Explore effectiveness of Reiki therapy as an adjuvant to conventional therapy in the management of stress and anxiety. Patients will be asked their stress level on a 1-10 scale before and after the Reiki intervention.
stress level: patient report | post intervention: immediately after Reiki
  Explore effectiveness of Reiki therapy as an adjuvant to conventional therapy in the management of stress and anxiety.

SECONDARY OUTCOMES:
salivary alpha amylase | baseline
  Examine whether a complementary therapy, such as Reiki, has any effect on the indices of physiological and subjective measurements when compared with the standard of care including nurse presence.
salivary alpha amylase | post intervention (after Reiki- 15 minutes from baseline)
  Examine whether a complementary therapy, such as Reiki, has any effect on the indices of physiological and subjective measurements when compared with the standard of care including nurse presence.
salivary alpha amylase | pre bone marrow biopsy (immediately before bone marrow is done, same day as Reiki)
  Examine whether a complementary therapy, such as Reiki, has any effect on the indices of physiological and subjective measurements when compared with the standard of care including nurse presence.
salivary alpha amylase | post bone marrow biopsy (immediately after bone marrow is done, same day as Reiki)
  Examine whether a complementary therapy, such as Reiki, has any effect on the indices of physiological and subjective measurements when compared with the standard of care including nurse presence.
salivary alpha amylase | 20 minutes post bone marrow biopsy
  Examine whether a complementary therapy, such as Reiki, has any effect on the indices of physiological and subjective measurements when compared with the standard of care including nurse presence.
salivary cortisol | baseline
  Examine whether a complementary therapy, such as Reiki, has any effect on the indices of physiological and subjective measurements when compared with the standard of care including nurse presence.
salivary cortisol | post intervention (after Reiki- 15 minutes from baseline)
  Examine whether a complementary therapy, such as Reiki, has any effect on the indices of physiological and subjective measurements when compared with the standard of care including nurse presence.
salivary cortisol | pre bone marrow biopsy (immediately before bone marrow is done, same day as Reiki)
  Examine whether a complementary therapy, such as Reiki, has any effect on the indices of physiological and subjective measurements when compared with the standard of care including nurse presence.
salivary cortisol | post bone marrow biopsy (immediately after bone marrow is done, same day as Reiki)
  Examine whether a complementary therapy, such as Reiki, has any effect on the indices of physiological and subjective measurements when compared with the standard of care including nurse presence.
salivary cortisol | 20 minutes post bone marrow biopsy
  Examine whether a complementary therapy, such as Reiki, has any effect on the indices of physiological and subjective measurements when compared with the standard of care including nurse presence.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Day, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States